CLINICAL TRIAL: NCT00093561
Title: Phase I Single Dose Pharmacokinetic Study of the Dietary Supplement Lycopene Delivered in Capsule Form to Healthy Male Volunteers Between 18 and 45 Years of Age
Brief Title: Lycopene in Preventing Prostate Cancer in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: UIC-2004-0040; CDR0000389223 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene

INTERVENTIONS:
Dietary Supplement: lycopene

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain substances to try to prevent the development or recurrence of cancer. The dietary supplement lycopene may prevent the development of prostate cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of lycopene in preventing prostate cancer in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and safety of lycopene supplementation as chemoprevention for prostate cancer in healthy participants.
* Determine the pharmacokinetics of this agent in these participants.
* Determine the dose range of this agent in these participants.

OUTLINE: This is a dose-escalation study.

Participants ingest a single-dose of oral lycopene over a maximum of 15 minutes on day 1.

Cohorts of 5 participants receive escalating doses of lycopene until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 participants experience dose-limiting toxicity.

Participants are evaluated periodically for 28 days.

PROJECTED ACCRUAL: A total of 25 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants in good medical condition

  * No chronic medical conditions
  * No regular use of prescription medications
  * No evidence of psychiatric disorder
  * Non-smoker

    * Former smokers allowed provided they have not smoked within the past 3 months
  * No history of alcohol abuse
* Serum lycopene concentration < 700 nM

PATIENT CHARACTERISTICS:

Age

* 18 to 45

Performance status

* Karnofsky 100%

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 13.0 g/dL
* WBC ≥ 4,000/mm^3
* Platelet count 150,000-400,000/mm^3

Hepatic

* AST and ALT ≤ 75 U/L
* Bilirubin ≤ 2.0 mg/dL
* No liver disease

Renal

* Creatinine ≤ 1.5 mg/dL
* No renal disease

Cardiovascular

* No cardiovascular disease
* No abnormal EKG

Other

* Within 15% of ideal body weight
* No history of gastrointestinal malabsorption or other condition that would preclude drug absorption
* No alcohol consumption within the past 72 hours
* No allergy to tomato-based products
* No history of cancer
* No diabetes mellitus
* No other illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 4 weeks since prior experimental drugs
* More than 14 days since prior prescription drugs
* No concurrent participation in another experimental trial
* No concurrent prescription drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2004-08; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Toxicity by blood chemistries and patient histories at 4 weeks after treatment
Pharmacokinetics by blood lycopene concentrations at 4 weeks after treatment

SECONDARY OUTCOMES:
Define dose range by blood lycopene concentrations at 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Rodvold, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Cancer Center, Chicago, Illinois, United States